CLINICAL TRIAL: NCT06930963
Title: The Influence of the Ankle-foot Orthoses on the Gross Motor Function of Children With Neurological Disorders
Brief Title: Impact of AFOs on the GMF of Children With CP or ABI
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: s65042
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Spastic Cerebral Palsy (sCP); Acquired Brain Injury
Keywords: Cerebral palsy; Gross motor function; Ankle-foot orthosis
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ambulatory children with CP or ABI: Ambulant children with cerebral palsy or acquired brain injury between 6 and 16 years old with a consistent gait pattern. They have prescribed ankle-foot orthoses by the medical team as part of the standard care.

SUMMARY:
Children with cerebral palsy (CP) or an acquired brain injury (ABI) are often prescribed ankle-foot orthoses (AFOs) to correct impairments of muscles and/or to prevent contractures and bony deformities. The impact of AFOs on gait, and to a lesser extent on gross motor function (GMF), has been investigated. Yet, little is known about their impact on the quality of movement. This study aims to examine how AFOs influence both the quality and capacity of daily functional activities in these children.

DETAILED DESCRIPTION:
Background:

Children with cerebral palsy (CP) or an acquired brain injury (ABI) often experience similar functional challenges and symptoms, leading to comparable treatment approaches. Enhancing gross motor function (GMF) and gait is a key treatment objective for children with CP or ABI, as these improvements are closely linked to functional independence and social participation. Ankle-foot orthoses (AFOs) are frequently prescribed to support gait, prevent secondary deformities, and compensate for muscle weakness. While existing research indicates that AFOs can enhance GMF capacity in children with CP, their impact on the quality of movement during functional tasks remains insufficiently explored.

Aim:

This study aims to evaluate the impact of AFOs on both the capacity (what children can do) and the quality (how they perform) of GMF in ambulatory children with CP or ABI. Specifically, the research seeks to determine the potential benefits or drawbacks of AFO use on specific functional tasks.

Methods/Study Design:

This prospective study will perform and film two GMFM-88-assessments (one with barefoot & one with AFOs) on 29 children with CP or ABI. Randomization to define the initial order of the assessment condition (barefoot or AFOs) will be performed by flipping a coin. Furthermore, these measurements will be performed with minimal 2 days and maximal 7 days in between and at similar moments during the day, representing an interval period that is sufficiently long (minimal 2 days) to minimalize possible test-potentiated learning effects and sufficiently short (maximal 7 days) to minimize potential impact of progression in functional skills due to rehabilitation sessions. The capacity of functional skills will be scored using the GMFM-88. The quality of the functional skills will be scored from the video of the GMFM-88 measurement, using the QFM. The videos of the two measurements will be scored separately with a minimal of 2 weeks in between, to minimize patient-specific performance expectations. An independent researcher will create two individual data sets of the recorded videos of the two GMFM-88 measurements (barefoot & AFO condition). The order in which the videos are divided over the two datasets, will be randomized.

The patients (with ABI or CP) will be recruited through the Cerebral Palsy Reference Center of the University Hospital (UZ) of Leuven (Prof. Dr. Anja Van Campenhout). Our preference goes to patients hospitalized in Pulderbos Revalidatiecentrum voor Kinderen en Jongeren or in UZ Leuven (Gasthuisberg), that are in their final phase of their intensive rehabilitation. Parents and children will be contacted by the involved researcher (Dra. Laure Everaert) via face-to-face conversation at the clinical appointment, via e-mail or by phone with the permission of the supervising medical doctor.

ELIGIBILITY:
Inclusion Criteria:

* Gross Motor Function Classification System (GMFCS) level I - III
* CP or ABI
* Age: 6 - 18 years
* Prescribed AFO by the medical team (as part of the standard care)

Exclusion Criteria:

* Severe contractures or spasticity, which makes it impossible to wear an AFO.
* Cognitive or visual impairment that limits the participation of the GMFM-88.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Ambulant children with cerebral palsy between 6 and 18 years old with a consistent gait pattern. They have prescribed ankle-foot orthoses by the medical team as part of the standard care.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
The GMFM-88 scores | Minimal 1 days and maximal 7 days between the two measurements and at similar moments during the day.
  Functional skill capacity will be assessed using the GMFM-88 in two conditions: once barefoot and once with AFOs.
The QFM scores | Minimal 1 days and maximal 7 days between the two measurements and at similar moments during the day.
  The quality of functional skills will be assessed using the QFM, based on video recordings of the GMFM-88 measurements under two conditions: once barefoot and once with AFOs.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, Prof. dr., Principal Investigator — Department of Rehabilitation Sciences, KU Leuven, Belgium
Locations (1):
- UZLeuven, Pellenberg, Belgium